CLINICAL TRIAL: NCT00162929
Title: A Phase I Study Investigating Multiple Injections of Autologous CD34+ Derived Dendritic Cells Transduced With an Adenovirus Expressing Rat Her-2/Neu in Patients With Metastatic or Locally Recurrent Breast Cancer
Brief Title: Her-2/Neu in Patients With Metastatic Breast Cancer (AdHERe)
Acronym: AdHERe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Cancer Research Network (Network); Canadian Breast Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTA-Control-092517
Record Dates: First submitted 2005-09-10; First posted 2005-09-13 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; locally recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: AdHer-2/neu transduced dendritic cells — Group 1 1 ×10'7 expanded cells (2.5 ×106 DCs per injection site) Group 2 5 ×10'7 expanded cells (1.25 ×107 DCs per injection site) Group 3 1 ×10'8 expanded cells (2.5 ×107 DCs per injection site)

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and/or maximum attainable dose of a vaccine consisting of human autologous dendritic cells transduced by an adenovector expressing rat Her-2/neu (AdHer-2/neu) in patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or locally recurrent breast cancer
2. 18 years of age or older
3. Her-2/neu positive (3+ by immunohistochemistry or fluorescence in-situ hybridization [FISH] +)
4. One of the following:

   1. currently receiving hormonal therapy or are candidates for such, or
   2. being considered for trastuzumab, or
   3. cancer has progressed on trastuzumab.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Prior or concurrent malignancies except for treated basal cell or squamous cell carcinoma of the skin or in situ cancer of the cervix or any other cancer treated and presumed cured for more than five years prior to study entry.
3. Currently receiving chemotherapy, immunotherapy, adenoviral gene therapy or biological cancer therapy. [Note: concurrent hormonal therapy (tamoxifen, aromatase inhibitors, or megace) is permitted.]
4. Treatment with trastuzumab within 4 weeks prior to first dose of vaccine therapy.
5. Hemoglobin < 80 g/L or granulocytes < 1.5 × 10^9/L or lymphocytes < 1.0 × 10^9/L or platelets < 100 × 10^9/L.
6. Baseline liver enzymes (AST or ALT) greater than 3 times the upper limit of normal or greater than 5 times the upper limit of normal if liver metastases are present and/or bilirubin is greater than 50 mmol.
7. CD4 cells < 0.5 ×10^9/L
8. Patients with documented brain metastases.
9. Patients with any acute illness that would interfere with the collection of CD34+ cells or administration of vaccination cellular therapy (i.e. unstable angina, renal or liver failure, or severe chronic obstructive airway disease).
10. Any patients requiring concurrent immunosuppressive therapy (e.g. corticosteroids).
11. Eastern Cooperative Oncology Group (ECOG) performance status of > 2.
12. Patients with a life expectancy of less than 6 months.
13. Geographic inaccessibility which would preclude follow-up. Patients registered on the trial must be treated and followed at the Juravinski Cancer Center and the Henderson site of the Hamilton Health Sciences.
14. Failure to give written informed consent.
15. Baseline left ventricular ejection fraction (LVEF) < 55% by echocardiography or multigated acquisition (MUGA) scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-01; Primary Completion 2009-07 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
toxicity | weeks 4, 6, 7, 10, 14, 18, 22, 26

SECONDARY OUTCOMES:
tumour response | Weeks 6, 18

CONTACTS AND LOCATIONS:
Overall Officials: Sukhbinder Dhesy-Thind, M.D., Study Chair — Ontario Clinical Oncology Group; Juravinski Cancer Centre - Hamilton Health Sciences; McMaster University; Ronan Foley, M.D., Principal Investigator — McMaster University; Richard Tozer, M.D., Principal Investigator — Juravinski Cancer Centre - Hamilton Health Sciences; Peter Ellis, M.D., Principal Investigator — Juravinski Cancer Centre - Hamilton Health Sciences; Jack Gauldie, M.D., Principal Investigator — McMaster University; Mark Levine, M.D., Principal Investigator — Ontario Clinical Oncology Group (OCOG)